CLINICAL TRIAL: NCT03076112
Title: Efficacy of Ipragliflozin Compared With Sitagliptin in Uncontrolled Type 2 Diabetes With Sulfonylurea and Metformin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Collaborators: Astellas Pharma Korea, Inc. (Industry)
Responsible Party: Principal Investigator, Soo Lim, Associate Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B-1612/375-004
Record Dates: First submitted 2017-03-06; First posted 2017-03-09 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Ipragliflozin; Sitagliptin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — ipragliflozin; Sitagliptin Phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ipragliflozin (Experimental): Ipragliflozin 50 mg in addition to their preexisting sulfonylurea and metformin
  ** Metformin and sulfonylurea's dosages
  * Metformin 500 mg - 2550 mg
  * Sulfonylurea: Glimepiride 1 mg - 8 mg or Gliclazide MR 30 mg - 120 mg
  Interventions: Drug: Ipragliflozin
- Sitagliptin (Active Comparator): Sitagliptin 100 mg in addition to their preexisting sulfonylurea and metformin
  ** Metformin and sulfonylurea's dosages
  * Metformin 500 mg - 2550 mg
  * Sulfonylurea: Glimepiride 1 mg - 8 mg or Gliclazide MR 30 mg - 120 mg
  Interventions: Drug: Sitagliptin

INTERVENTIONS:
Drug: Ipragliflozin — Ipragliflozin as add-on to Metformin and Sulfonylurea in patients with poorly controlled type 2 diabetes
  Other Names: Suglat
  Arms: Ipragliflozin
Drug: Sitagliptin — Sitagliptin as add-on to Metformin and Sulfonylurea in patients with poorly controlled type 2 diabetes
  Other Names: Januvia
  Arms: Sitagliptin

SUMMARY:
The objectives of this study are 1) to compare the effect of ipragliflozin 50 mg on glucose-lowering effect with sitagliptin 100 mg in patients with type 2 diabetes mellitus, whose HbA1c level is ≥ 7.5% with sulfonylurea and metformin, 2) to investigate changes of other metabolic and cardiovascular risk factors such as triglyceride, HDL-cholesterol, uric acid, blood pressure, and inflammatory markers, 3) to examine changes of body composition including fat and muscle mass with volume status.

DETAILED DESCRIPTION:
The objectives of this study are to compare the effect of 50mg of ipragliflozin, a SGLT2 inhibitor, on glucose-lowering effect with 100mg of sitagliptin, a DPP4 inhibitor in patients with type 2 diabetes mellitus, whose HbA1c level is ≥ 7.5% with sulfonylurea and metformin.

We are also going to investigate changes of other metabolic and cardiovascular risk factors such as triglyceride, HDL-cholesterol, uric acid, blood pressure, and inflammatory markers.

Changes of body composition including fat and muscle mass with volume status will be also examined.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes with HbA1c 7.5% - 9.0% at screening visit
* Male or female between 20 and 75 years of age
* Patients taking sulfonylurea (glimepiride 1~8mg or gliclazide 30~120 mg or equivalent dose) and metformin (≥ 1000 mg or maximum tolerated dose) for more than 3 months
* BMI ≥23 kg/m²
* Estimated GFR ≥ 60 ml/min/1.73m²
* Women of child bearing potential must take precautions to avoid pregnancy throughout the study and for 4 weeks after intake of the last dose and must have a negative urinary pregnancy test.

Exclusion Criteria:

* Type 1 diabetes, gestational diabetes, or diabetes with secondary cause
* Patients with acute coronary syndrome within 3 months prior to screening visit
* Patients with acute coronary syndrome within 3 months prior to screening visit
* Pregnant or breastfeeding women or reproductive-age women who refuse contraception
* Chronic hepatitis B or C (except healthy carrier of HBV), liver disease (AST/ALT > 3-fold the upper limit of normal)
* Cancer within 5 years (except squamous cell cancer, cervical cancer, thyroid cancer with appropriate treatment) except thyroid cancer or carcinoma in situ
* Other clinical trials within 30 days
* Alcohol abuse
* Contraindication to SGLT2 inhibitors or Dipeptidyl-peptidase 4 inhibitors
* Taking insulin, oral hypoglycemic agents other than metformin, sulfonylurea, and the study drugs.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2017-04-25 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Glycated hemoglobin | Baseline, week 12, week 24
  Change of HbA1c after 24 weeks' treatment

SECONDARY OUTCOMES:
Glycemic target goal achievement | Baseline, week 12, week 24
  Glycemic target goal achievement (HbA1c < 7%) at week 24
Body weight | Baseline, week 12, week 24
  Change of body weight at week 24
Body fat mass | Baseline, week 24
  Change of body fat mass at week 24
Fasting plasma glucose level | Baseline, week 12, week 24
  Change of fasting plasma glucose level at week 24
Postprandial 2hr glucose level | Baseline, week 12, week 24
  Changes of postprandial 2hr glucose level at week 24
Blood Pressure | Baseline, week 12, week 24
  Change of systolic/diastolic blood pressure at week 24
Triglyceride/HDL-cholesterol ratio | Baseline, week 12, week 24
  Changes of triglyceride/HDL-cholesterol ratio at week 24
Uric acid | Baseline, week 12, week 24
  Changes of uric acid at week 24
Parathyroid hormone | Baseline, week 12, week 24
  Changes of parathyroid hormone at week 24
25-hydroxyvitamin D | Baseline, week 12, week 24
  Changes of 25-hydroxyvitamin D at week 24

CONTACTS AND LOCATIONS:
Overall Officials: Soo Lim, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
Yes

REFERENCES:
- [Background] Hedrington MS, Davis SN. Ipragliflozin , a sodium-glucose cotransporter 2 inhibitor, in the treatment of type 2 diabetes. Expert Opin Drug Metab Toxicol. 2015 Apr;11(4):613-23. doi: 10.1517/17425255.2015.1009893. Epub 2015 Feb 2. PMID 25643044
- [Background] Kadokura T, Zhang W, Krauwinkel W, Leeflang S, Keirns J, Taniuchi Y, Nakajo I, Smulders R. Clinical pharmacokinetics and pharmacodynamics of the novel SGLT2 inhibitor ipragliflozin. Clin Pharmacokinet. 2014 Nov;53(11):975-88. doi: 10.1007/s40262-014-0180-z. PMID 25316572
- [Background] Veltkamp SA, van Dijk J, Collins C, van Bruijnsvoort M, Kadokura T, Smulders RA. Combination treatment with ipragliflozin and metformin: a randomized, double-blind, placebo-controlled study in patients with type 2 diabetes mellitus. Clin Ther. 2012 Aug;34(8):1761-71. doi: 10.1016/j.clinthera.2012.06.027. Epub 2012 Jul 15. PMID 22795925
- [Background] Takasu T, Hayashizaki Y, Tahara A, Kurosaki E, Takakura S. Antihyperglycemic effect of ipragliflozin, a sodium-glucose co-transporter 2 inhibitor, in combination with oral antidiabetic drugs in mice. Clin Exp Pharmacol Physiol. 2015 Jan;42(1):87-93. doi: 10.1111/1440-1681.12317. PMID 25311502
- [Background] Smulders RA, Zhang W, Veltkamp SA, van Dijk J, Krauwinkel WJ, Keirns J, Kadokura T. No pharmacokinetic interaction between ipragliflozin and sitagliptin, pioglitazone, or glimepiride in healthy subjects. Diabetes Obes Metab. 2012 Oct;14(10):937-43. doi: 10.1111/j.1463-1326.2012.01624.x. Epub 2012 Jun 7. PMID 22587345
- [Background] Macdonald FR, Peel JE, Jones HB, Mayers RM, Westgate L, Whaley JM, Poucher SM. The novel sodium glucose transporter 2 inhibitor dapagliflozin sustains pancreatic function and preserves islet morphology in obese, diabetic rats. Diabetes Obes Metab. 2010 Nov;12(11):1004-12. doi: 10.1111/j.1463-1326.2010.01291.x. PMID 20880347
- [Background] Bolinder J, Ljunggren O, Johansson L, Wilding J, Langkilde AM, Sjostrom CD, Sugg J, Parikh S. Dapagliflozin maintains glycaemic control while reducing weight and body fat mass over 2 years in patients with type 2 diabetes mellitus inadequately controlled on metformin. Diabetes Obes Metab. 2014 Feb;16(2):159-69. doi: 10.1111/dom.12189. Epub 2013 Aug 29. PMID 23906445
- [Background] Matthaei S, Bowering K, Rohwedder K, Grohl A, Parikh S; Study 05 Group. Dapagliflozin improves glycemic control and reduces body weight as add-on therapy to metformin plus sulfonylurea: a 24-week randomized, double-blind clinical trial. Diabetes Care. 2015 Mar;38(3):365-72. doi: 10.2337/dc14-0666. Epub 2015 Jan 15. PMID 25592197
- [Background] Hermansen K, Kipnes M, Luo E, Fanurik D, Khatami H, Stein P; Sitagliptin Study 035 Group. Efficacy and safety of the dipeptidyl peptidase-4 inhibitor, sitagliptin, in patients with type 2 diabetes mellitus inadequately controlled on glimepiride alone or on glimepiride and metformin. Diabetes Obes Metab. 2007 Sep;9(5):733-45. doi: 10.1111/j.1463-1326.2007.00744.x. Epub 2007 Jun 26. PMID 17593236